CLINICAL TRIAL: NCT00041860
Title: Modulation of Benzene Metabolism by Exposure to Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 9676-CP-001
Record Dates: First submitted 2002-07-18; First posted 2002-07-22 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-07

CONDITIONS: Lung Diseases; Cancer
Keywords: Benzene; Air pollution
MeSH Terms: conditions — Lung Diseases; Neoplasms

INTERVENTIONS:
Procedure: Controlled Exposure to Environmental Contaminant

SUMMARY:
The research is to evaluate benzene metabolism after exposure at levels that can be found in the environment, such as the higher end concentrations in the air inside cars and buses while being driven in heavy traffic and inside private and public parking garages. To do so breath, urine, and blood samples prior to, during and after being exposed to benzene as well as benzene levels and benzene metabolites present are measured.

DETAILED DESCRIPTION:
The research is to evaluate benzene metabolism after exposure at levels that can be found in the environment, such as the higher end concentrations in the air inside cars and buses while being driven in heavy traffic and inside private and public parking garages. To do so breath, urine, and blood samples prior to, during and after being exposed to benzene as well as benzene levels and benzene metabolites present are measured. The exposures take place in the Controlled Environmental Facility operated by the Environmental and Occupational Health Sciences Institute (EOHSI). This allows us to control the exact benzene air level and to use benzene containing 13C, a stable (non-radioactive) form of carbon, one of the atoms that make up benzene. Isotopes are different forms of the same atom. Using 13C will allow us to tell the difference between the benzene and the compounds it changes to in the body that come from our experiment compared to what is present in your body from other sources. In addition to just benzene exposure on some days the subject is also be exposed to methyl tertiary butyl ether (MTBE), another component of gasoline, to take an iron supplement pill and/or to take vitamins C and E pills. How benzene is metabolized or changed in the body will be compared for these differences to better understand how the body deals with benzene.

Age Groups: Child, Adult, Older Adult